CLINICAL TRIAL: NCT00371865
Title: Acceptance-Based Treatment for Chronic Pain
Brief Title: Behavioral Treatments for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F4306-I
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Intractable Pain
Keywords: Behavior therapy; Chronic pain; Cognitive therapy; Meditation; Mindfulness; Psychotherapy
MeSH Terms: conditions — Pain, Intractable; Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (Active Comparator): 8 group-administered sessions of Cognitive-Behavioral Therapy
  Interventions: Behavioral: Cognitive-behavioral therapy
- Acceptance-Based Therapy (Experimental): 8 group-administered sessions of Acceptance-based therapy
  Interventions: Behavioral: Acceptance-based therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — 8 group-administered sessions of Cognitive-Behavioral Therapy; includes relaxation, cognitive restructuring, and problem-solving
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy
Behavioral: Acceptance-based therapy — 8 group-administered sessions of Acceptance-based therapy; includes mindfulness, values, and committed action
  Other Names: ACT
  Arms: Acceptance-Based Therapy

SUMMARY:
The purpose of the study is to test a brief, group-administered psychosocial intervention to reduce interference of pain with daily life, emotional distress, and pain intensity, and improve quality of life and physical activity levels in individuals with chronic pain.

DETAILED DESCRIPTION:
Chronic pain affects at least 15% of the veteran population and represents a high priority for the VA. In addition to primary pain conditions, chronic pain is a common secondary condition resulting from battlefield injuries, traumatic accidents, and congenital and acquired disorders. Unlike most forms of acute pain, treatment options available for patients suffering from chronic pain frequently offer only short-term or partial relief from symptoms. The focus of rehabilitative intervention thus becomes the reduction of disability and emotional distress and improvement in quality of life and activity levels.

Chronic pain rehabilitation has evolved from a primarily one-dimensional, medically oriented approach to a multidisciplinary approach that incorporates a biopsychosocial formulation to pain management with physiological, cognitive, behavioral, and emotional components. This conceptualization of pain recognizes that multiple intervention modalities, including psychosocial approaches, are required when providing treatment to chronic pain patients.

A relatively new psychosocial approach to chronic pain management and rehabilitation involves acceptance of pain-related experiences. The Acceptance-based Therapy (AT) model is based on the theory that attempts to escape, avoid, or control negative experiences that cannot be changed, such as chronic pain, may paradoxically contribute to the increased experience of them. Instead of seeking to control the negative experience, AT teaches individuals to use mindfulness strategies to enlarge the scope of experience beyond pain and to engage in behaviors that are consistent with personal values and goals when total elimination of pain or other negative experiences is not possible. Empirical support for acceptance-based approaches to chronic pain management is growing. Data from one of the first comparisons of AT to a well-established psychosocial intervention, Cognitive-Behavioral Therapy (CBT), performed at VASDHS by the PI, suggests that AT may be superior to CBT as an adjunctive treatment for chronic pain.

The proposed study assembles a multidisciplinary team with extensive experience in chronic pain interventions research to evaluate the benefits of a brief, manualized group-administered psychosocial intervention which could be easily integrated into multidisciplinary pain rehabilitation programs throughout the VA system to reduce disability in veterans with chronic pain secondary to other conditions. Specifically, we propose to examine the effects of a promising new chronic pain intervention based on AT principles on the primary outcome of pain interference and secondary outcomes of emotional distress, quality of life, physical activity, pain intensity, and treatment satisfaction among 94 veterans with chronic benign pain as a secondary condition. The AT intervention will be compared with treatment as usual (TAU) in a within-subjects design and with CBT in a randomized, between-subjects design. Outcomes include an objective measure of physical activity, actigraphy, as well as self-reported measures and will be evaluated at baseline, 6 weeks (after a TAU phase), 12 weeks (after treatment), and at a 6-month follow-up period to investigate maintenance of gains. The study design also allows for an investigation of hypothesized mechanisms of change, acceptance (for AT) and perceived pain control (for CBT). Thus, the proposed project has the potential to enhance the current VA standard of care as well as to add to the scientific literature on psychological models and rehabilitation of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older;
* Proficient in English;
* Willing and able to provide written informed consent (proposed informed consent form attached as Appendix A);
* Diagnosis of chronic benign pain as a secondary condition associated with a primary impairment due to a traumatic injury or congenital or acquired disorder as verified by a study physician after a medical diagnostic evaluation;
* Average pain severity rated > 4/10 with resulting functional limitations; and
* Pain duration of at least 6 months.

Exclusion Criteria:

* Participation in psychotherapy for pain the past 2 months;
* Serious, unstable medical illness for which inpatient hospitalization is likely over the next 3 months; and
* The following DSM-IV diagnoses or active problems within the past 6 months noted in the patient's CPRS medical record or diagnosed during a structured psychiatric interview: 1) schizophrenia; 2) other psychotic disorder; 3) bipolar disorder; 4) organic mental disorder; 5) borderline or antisocial personality disorder; or 6) alcohol or substance abuse or dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Wetherell, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

REFERENCES:
- [Result] Wetherell JL, Afari N, Rutledge T, Sorrell JT, Stoddard JA, Petkus AJ, Solomon BC, Lehman DH, Liu L, Lang AJ, Atkinson HJ. A randomized, controlled trial of acceptance and commitment therapy and cognitive-behavioral therapy for chronic pain. Pain. 2011 Sep;152(9):2098-2107. doi: 10.1016/j.pain.2011.05.016. Epub 2011 Jun 17. PMID 21683527
- [Result] Mostoufi SM, Afari N, Ahumada SM, Reis V, Wetherell JL. Health and distress predictors of heart rate variability in fibromyalgia and other forms of chronic pain. J Psychosom Res. 2012 Jan;72(1):39-44. doi: 10.1016/j.jpsychores.2011.05.007. Epub 2011 Jun 30. PMID 22200521

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy | Acceptance-Based Therapy
Started | 57 | 57
Completed | 42 (7 withdrew before starting the intervention. 8 withdrew after starting the intervention.) | 43 (8 withdrew before starting the intervention. 6 withdrew after starting the intervention.)
Not Completed | 15 | 14
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy | Acceptance-Based Therapy | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (12.5) | 54.9 (12.5) | 54.9 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 28 | 28 | 56
Race/Ethnicity, Customized [Number; unit: participants]
  NonHispanic white | 38 | 39 | 77
  Other | 19 | 18 | 37
Region of Enrollment [Number; unit: participants]
  United States | 57 | 57 | 114

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory
Description: This questionnaire measures pain severity and interference. Scores range from 0-10, with higher scores indicating more pain.
Time Frame: 12 weeks (post treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: 8 group-administered sessions of Cognitive-Behavioral Therapy
  Cognitive-behavioral therapy: 8 group-administered sessions of Cognitive-Behavioral Therapy; includes relaxation, cognitive restructuring, and problem-solving
- Arm 2: 8 group-administered sessions of Acceptance-based therapy
  Acceptance-based therapy: 8 group-administered sessions of Acceptance-based therapy; includes mindfulness, values, and committed action
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 57 | 57
units on a scale | 4.5 (2.7) | 5.1 (2.4)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = .27, Mixed Models Analysis

2. Secondary Outcome: West Haven-Yale Multidimensional Pain Inventory - Activity Subscales
Description: This questionnaire measures levels of activity that can be affected by pain. Full measure has a range of 0-6, with higher scores indicating higher levels of activity.
Time Frame: 12 weeks (post treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 57 | 57
units on a scale | 2.3 (0.8) | 2.0 (0.8)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = .90, Mixed Models Analysis

3. Secondary Outcome: SF-12
Description: This questionnaire measures quality of life. Scores range from 0 to 100, with higher scores indicating better quality of life.
Time Frame: 12 weeks (post treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 57 | 57
units on a scale | 44.9 (12.1) | 41.0 (13.6)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = .13, Mixed Models Analysis

4. Secondary Outcome: Beck Depression Inventory
Description: This questionnaire measures depressive symptoms. Scores range from 0 to 63, with higher scores indicating higher levels of depressive symptoms.
Time Frame: 12 weeks (post treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 57 | 57
units on a scale | 13.2 (11.1) | 17.8 (12.2)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = .26, Mixed Models Analysis

5. Secondary Outcome: Pain Anxiety Symptom Scale - 20
Description: This questionnaire measures pain-related anxiety. Scores range from 0 to 100, with higher scores indicating higher levels of anxiety.
Time Frame: 12 weeks (post treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 57 | 57
units on a scale | 37.9 (20.7) | 41.5 (23.4)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = .90, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No